CLINICAL TRIAL: NCT00040833
Title: Acupuncture for the Treatment of Pancreatic Cancer Pain: A Single Arm Phase II Study
Brief Title: Acupuncture and Acupressure in Treating Patients With Moderate or Severe Pain Related to Stage III or Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: 02-008; CDR0000069411 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2082
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Pain; Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; pain; stage IV pancreatic cancer
MeSH Terms: conditions — Pain; Pancreatic Neoplasms | interventions — Analgesia

INTERVENTIONS:
Procedure: complementary or alternative medicine procedure
Procedure: pain therapy

SUMMARY:
RATIONALE: Acupuncture and acupressure may help relieve moderate or severe pain associated with stage III or stage IV pancreatic cancer.

PURPOSE: Phase II trial to study the effectiveness of acupuncture and accupressure in treating patients who have moderate or severe pain associated with stage III or stage IV pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the effects of acupuncture and acupressure on pain, sedation, and use of opiate medication in patients with moderate or severe pain related to stage III or IV pancreatic cancer.
* Determine whether controlled trials of this therapy are warranted in this patient population.
* Provide data to aid design of further warranted studies of this therapy in this patient population.

OUTLINE: Patients receive acupuncture treatment comprising 20 minutes of needle insertion into the arms and abdomen to the depth used in traditional Chinese medicine on approximately days 4, 7, 11, and 14. After each acupuncture treatment, the acupuncturist applies/reapplies acupressure devices by inserting 2-6 smaller needles (studs) into the abdomen (which are held in place with surgical tape) and taping tiny metal balls to 3 points in each ear. Patients or caregivers are instructed to administer acupressure by pressing on the ear points (metal balls) for 1-2 minutes per point and moving the semi-permanent abdominal needles in small circular movements with the fingers, at a rate of 2-3 cycles per second, for 1-2 minutes per point, upon waking in the morning and in the early afternoon. Patients or caregivers are also instructed to stimulate a "rescue point" (the Shenmen auricular point) if patients experience pain exacerbations at other times during the day. Patients who respond well to acupuncture are offered further treatment.

Pain is assessed using the numerical rating scale on approximately days 1-4, 7, 11, and 14-17. Sedation is assessed using the Profile of Mood States (POMS) on approximately days 3 and 17. Analgesic medication use is assessed on approximately days 1-3 and 15-17.

PROJECTED ACCRUAL: A total of 10-29 patients will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage III or IV primary pancreatic cancer
* At least 4 days since prior change in type of pain medication
* No change in dose of long-acting analgesics
* Actual dose of as needed (PRN) pain medication may vary
* One of the following pain scores:

  * Pain score of at least 4 on a scale of 0 to 10
  * A score of at least 54 out of 88 on the combined relevant Profile of Mood States (POMS) subscales (Vigor, Fatigue, and Confusion) with no evidence that sedation results from cause other than opiate medication and patient reported using PRN opiates on at least 4 of the past 7 days (patients who are eligible for this study on the basis of POMS scores must be taking PRN medication)

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Not specified

Life expectancy:

* At least 4 weeks

Hematopoietic:

* Absolute neutrophil count at least 500/mm^3
* Platelet count at least 20,000/mm^3

Hepatic:

* INR no greater than 2.5

Renal:

* Not specified

Cardiovascular:

* No heart valve dysfunction

Other:

* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior gemcitabine unless there is documented disease progression
* Concurrent chemotherapy (except gemcitabine) allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 1 week since prior epidural analgesia, celiac plexus block, or thoracoscopic or open splanchnicectomy
* No concurrent epidural analgesia, celiac plexus block, or thoracoscopic or open splanchnicectomy

Other:

* See Disease Characteristics
* At least 3 months since prior acupuncture
* Concurrent experimental treatments allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barrie R. Cassileth, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States